CLINICAL TRIAL: NCT03843242
Title: Evaluation of Ventricular Pacing Suppression Algorithms in Dual Chamber
Brief Title: Evaluation of Ventricular Pacing Suppression Algorithms in Dual Chamber Pacemaker
Acronym: LEADER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Principal Investigator, Seongwook Han, Professor of Internal Medicine, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018-08-022
Record Dates: First submitted 2019-02-11; First posted 2019-02-18 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Sick Sinus Syndrome; Pacemaker; Heart Failure
MeSH Terms: conditions — Sick Sinus Syndrome; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pacemaker with Fixed long AV delay (Experimental): 1. Patients who meet the inclusion criteria and is implanted with a Biotronik Enitra 8 DR-T pacemaker are eligible.
  2. The pacemaker was programmed with a long and fixed atrioventricular interval for the first 3 months.
  3. Definition of fixed AV delay (than intrinsic AV conduction) • If P-wave exists: intrinsic AV conduction time = As ~ Vs interval in the marker channel sensed AV delay = intrinsic AV conduction time + 20 msec paced AV delay = sensed AV delay + 30 msec • If no P-wave exits: intrinsic AV conduction time = Ap ~ Vs interval in the marker channel paced AV delay = intrinsic AV conduction time + 20 msec sensed AV delay = paced AV delay - 30 msec • If the intrinsic AV conduction time is ≥ 300ms, make paced/sensed AV delay 350/320 msec
  Interventions: Device: Pacemaker with Fixed long AV delay
- Pacemaker with VpS® algorithm on (Experimental): Vp Suppression ON algorithm: This feature promotes the intrinsic AV conduction by only pacing the ventricle when intrinsic conduction becomes unstable or disappears. Depending on the presence or absence of AV conduction, the feature is implemented either in the ventricular pacing suppression state ADI(R), which promotes the intrinsic conduction, or in the DDD(R) ventricular pacing state Vp DDD(R), which provides ventricular pacing. Automatic switching capabilities between those two states promotethe intrinsic conduction as much as possible without harming the patient. Scheduled Vs searching tests look for intrinsic conduction using an extended AV delay of 450ms.
  Interventions: Device: Pacemaker with Fixed long AV delay; Device: Pacemaker with VpS® algorithm on
- Pacemaker with IRSplus algorithm on (Experimental): IRS plus algorithm: This algorithm incorporates two different functions: the first is scan hysteresis, which better enables the heart to pace on its own by periodically extending the search time for its natural pacing stimulus (the intrinsic AV conduction) over six consecutive atrial cycles. The second is the repetitive hysteresis, which recognizes when the heart is not pacing on its own (a consistent loss of intrinsic AV conduction lasting for six consecutive atrial cycles) and switches the mode of the device from extended to basic atrioventricular (AV) delay.
  Interventions: Device: Pacemaker with Fixed long AV delay; Device: Pacemaker with IRSplus algorithm on

INTERVENTIONS:
Device: Pacemaker with Fixed long AV delay — Fixed AV delay was applied in the first 3 months of pacemaker implantation according to previously proposed definition.
Device: Pacemaker with VpS® algorithm on — 1. After first 3 months of pacemaker implantation, the patients will be randomized into two groups (Vp-suppression algorithm on group vs. IRS-plus algorithm on group) using a centralized randomization system.
  2. In Vp-suppression algorhithm on group, Vp suppression algorithm of Enitra 8 DR-T pacemaker will be turned on at 3month visit after enrollment.
  3. The patient will be followed at 3-month after enrollment and at 6-month and 12-month after applying the specific algorithm.
  Arms: Pacemaker with VpS® algorithm on
Device: Pacemaker with IRSplus algorithm on — 1. After first 3 months of pacemaker implantation, the patients will be randomized into two groups (Vp-suppression algorithm on group vs. IRS-plus algorithm on group) using a centralized randomization system.
  2. In IRS-plus algorithm on group, IRS plus algorithm of Enitra 8 DR-T pacemaker will be turned on at 3 month visit after enrollment.
  3. The patient will be followed at 3-month after enrollment and at 6-month and 12-month after applying the specific algorithm.
  Arms: Pacemaker with IRSplus algorithm on

SUMMARY:
The recent study using IRSplus and VpS algorithm from Biotronik pacemaker showed the significant reduction in ventricular pacing to less than 3%.

The purpose of this study is to evaluate the efficacy of IRSplus and VpS algorithm in reducing ventricular pacing compared with conventional DDD pacing with a fixed AV delay.

DETAILED DESCRIPTION:
The adverse cardiac outcomes due to right ventricular apical pacing with dual chamber pacemakers have been widely observed such as ventricular dyssynchrony resulting in reduced left ventricular function, increased risk of heart failure and atrial fibrillation. To minimize the ventricular pacing, manufacturers of pacemaker have made an effort to develop special algorithms designed to deliver right ventricular pacing only in case of demonstrated persistent long PR interval or repetitively lacking intrinsic ventricular activation.

Currently, there are three methods and algorithms are available with a pacemaker from the Biotronik SE & Co. KG to minimize right ventricular pacing as follows; DDD mode with fixed longer atrioventricular (AV) delay than intrinsic conduction time; Intrinsic rhythm support (IRSplus); Ventricular pacing suppression (VpS).

In the real world, it is the most common practice to program the DDD(R) mode with fixed long AV delay because of physician's concerns about the possible failure of an algorithm or long pause being resulted from 2 consecutive loss of AV conduction by the algorithm. However, the main disadvantage of a fixed with long AV delay is that the prolonged total atrial refractory period (TARP) results in changes of the upper rate behavior (i.e., pseudo-Wenckebach AV block and subsequently 2:1 block at lower atrial tracking rates). The possibility of pacemaker-mediated tachycardia is getting high if the post-ventricular atrial refractory period (PVARP) is shortened to compensate. Furthermore, there is a high chance to have fusion/pseudo-fusion of ventricular pacing in a fixed long AV delay because the AV conduction is dynamic according to the heart rate.

The recent systematic review showed that there are no significant differences between the pacing modes for mortality, heart failure, stroke, and atrial fibrillation (AF) in patients with sinus node dysfunction (SND) without AV block. However, the dual chamber pacemaker is still recommended in patients with SND due to lack of tools to identify patients at high risk of developing the complete AV block. The meta-analysis about the effect of the reduction in unnecessary ventricular pacing using a sophisticated algorithm in patients with SND showed there are no benefits in clinical outcomes compared with conventional DDD mode. But the percentage of ventricular pacing in ventricular pacing reduction modality group was not negligible between 1~11.5%. The result might be changed if we have data with a more significant reduction in ventricular pacing using difference algorithm. The recent study using IRSplus and VpS algorithm from Biotronik pacemaker showed the significant reduction in ventricular pacing to less than 3%.

The purpose of this study is to evaluate the efficacy of IRSplus and VpS algorithm compared with conventional DDD pacing with a fixed AV delay.

ELIGIBILITY:
Inclusion Criteria:

* Sick sinus syndrome
* No evidence of 2nd and 3rd degree AV block
* Provide written informed consent
* Age ≥ 20 years old

Exclusion Criteria:

* 2nd and 3rd degree AV block
* History of AF
* patients with older version of pacemaker
* Life expectancy ≤ one year
* Pregnant or lactating women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Percentage of right ventricular pacing | During first 3 months after the study enrollment
  the right ventricle pacing percentage appeared on the pacemaker interrogation
Percentage of right ventricular pacing | During 4 ~ 9 months after the study enrollment
  the right ventricle pacing percentage appeared on the pacemaker interrogation
Percentage of right ventricular pacing | During 10 ~ 15 months after the study enrollment
  the right ventricle pacing percentage appeared on the pacemaker interrogation

SECONDARY OUTCOMES:
New onset atrial fibrillation | During 12 months after randomization (15 months after enrollment)
  Percentage of patients with new onset atrial fibrillation during the observation period
Occurrence of heart failure | During 12 months after randomization (15 months after enrollment)
  Percentage of patients who experienced symptomatic heart failure during the observation period
Percentage of atrial high rate episode | During 12 months after randomization (15 months after enrollment)
  Percentage of atrial high rate episode appeared on the pacemaker interrogation

CONTACTS AND LOCATIONS:
Overall Officials: Seongwook Han, M.D., Ph.D., Study Chair — Keimyung University Dongsan Medical Center
Locations (6):
- South Korea (6):
  - Daegu Fatima Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Kyungpook National University Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Yeungnam University Hospital, Daegu
  - Division of Cardiology, Department of Internal Medicine, Daegu Catholic University Medical Center, Daegu
  - Dongguk University Medical Center, Ilsan
  - Pusan National University Hospital, Pusan